CLINICAL TRIAL: NCT00360282
Title: Effect of Rizatriptan on Rotational Motion Sickness in Migraineurs
Brief Title: Does a Migraine Medication Decrease Rotational Motion Sickness in People Suffering From Migraines?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Joseph Furman, Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 0602009; 31449 (Other: Merck)
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Migraine
Keywords: Migraine; Triptans; Motion Sickness
MeSH Terms: conditions — Migraine Disorders; Motion Sickness | interventions — rizatriptan; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- With Vertigo; Placebo - Rizatriptan (Other): This group received placebo on visit 1 and Rizatriptan on visit 2.
  Interventions: Drug: Rizatriptan; Other: Placebo
- With Vertigo; Rizatriptan - Placebo (Other): These subjects received Rizatriptan on visit 1 and placebo on visit 2.
  Interventions: Drug: Rizatriptan; Other: Placebo
- Without Vertigo; Placebo - Rizatriptan (Other): This group received placebo on visit 1 and Rizatriptan on visit 2.
  Interventions: Drug: Rizatriptan; Other: Placebo
- Without Vertigo; Rizatriptan-Placebo (Other): This group received Rizatriptan on visit 1 and placebo on visit 2.
  Interventions: Drug: Rizatriptan; Other: Placebo

INTERVENTIONS:
Drug: Rizatriptan — 10 mg Rizatriptan in an unlabeled pill given once on one of two visits
  Other Names: Maxalt
Other: Placebo — In an unlabeled pill given once on one of two visits.
  Other Names: Sugar Pill

SUMMARY:
The purpose of this study is to determine if Rizatriptan, a migraine medication, lowers motion sickness in migraine sufferers.

DETAILED DESCRIPTION:
Migraine sufferers undergo vestibular tests and were excluded if there were clinically significant abnormalities. Following screening, there were 2 experimental visits in which migraine sufferers were pre-treated with either Rizatriptan or placebo. After taking the drug, subjects were idle for 2 hours. Baseline motion sickness and subjective units of distress levels were assessed prior to undergoing sinusoidal-earth-vertical earth axis rotation in darkness at 0.05 Hz. Scores were taken immediately after stopping. Subjects were given a 2 minutes rest and then underwent a motion sickness provoking rotation. Subjective scores were assessed immediately following. Another two minute rest was given and if the subject was able, underwent a second motion sickness provoking stimulus followed by an assessment.

ELIGIBILITY:
Inclusion Criteria:

* History of motion sickness
* Currently suffering from migraines with at least 2 episodes during the previous 12 months
* Previous use and tolerance to triptans

Exclusion Criteria:

* Current tobacco user
* History of or current hypertension, cardiac disease, arrhythmia, hypercholesterolemia, hemiplegic/basilar migraine, stroke, diabetes, vascular disease or kidney disease
* Family history of early myocardial infarction (first-degree relative < 45 years old at time of event)
* Constant dizziness or constant vestibular symptoms
* History of ear, nose and throat (ENT) disease, e.g. Meniere's disease
* Current treatment with propranolol or medications that would preclude use of a triptan(e.g. ergotamine)
* Major vestibular abnormality found on screening
* Testing positive on over-the-counter pregnancy test
* Taken an Monamine Oxidase (MAO) inhibitor within two weeks of testing
* Allergy or intolerance to gelatin
* Corrected visual acuity of > 20/40 O.U.
* Women who are pregnant or breastfeeding

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Furman, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Furman JM, Marcus DA, Balaban CD. Rizatriptan reduces vestibular-induced motion sickness in migraineurs. J Headache Pain. 2011 Feb;12(1):81-8. doi: 10.1007/s10194-010-0250-z. Epub 2010 Sep 23. PMID 20862509
- [Derived] Webster KE, Dor A, Galbraith K, Haj Kassem L, Harrington-Benton NA, Judd O, Kaski D, Maarsingh OR, MacKeith S, Ray J, Van Vugt VA, Burton MJ. Pharmacological interventions for acute attacks of vestibular migraine. Cochrane Database Syst Rev. 2023 Apr 12;4(4):CD015322. doi: 10.1002/14651858.CD015322.pub2. PMID 37042545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the general public in Pittsburgh, PA from October 2006 until November 2008.
Pre-assignment Details: 36 subjects recruited; 9 were not assigned to a group (3 did not not meet migraine inclusion criteria, 1 was excluded on vestibular screening results, 1 withdrew, 4 were lost to follow up)
Groups:
- With Vertigo; Placebo-Rizatriptan: These participants suffered from migraines with associated dizziness/vertigo. They were given placebo on visit one and Rizatriptan on visit 2.
- Without Vertigo; Placebo - Rizatriptan: These participants suffered from migraines but did not have associated dizziness/vertigo. This group received placebo on visit 1 and Rizatriptan on visit 2.
- With Vertigo; Rizatriptan - Placebo: These participants suffered from migraine and had associated vertigo/dizziness. They received Rizatriptan on visit 1 and placebo on visit 2.
- Without Vertigo; Rizatriptan - Placebo: These participants suffered from migraine without associated vertigo/dizziness. They received Rizatriptan on visit 1 and placebo on visit 2.
Period: First Intervention
Arm/Group | With Vertigo; Placebo-Rizatriptan | Without Vertigo; Placebo - Rizatriptan | With Vertigo; Rizatriptan - Placebo | Without Vertigo; Rizatriptan - Placebo
Started | 6 | 8 | 7 | 6
Completed | 6 | 8 | 7 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Washout 1-3 Weeks
Arm/Group | With Vertigo; Placebo-Rizatriptan | Without Vertigo; Placebo - Rizatriptan | With Vertigo; Rizatriptan - Placebo | Without Vertigo; Rizatriptan - Placebo
Started | 6 | 8 | 7 | 6
Completed | 6 | 8 | 6 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Period: Second Intervention
Arm/Group | With Vertigo; Placebo-Rizatriptan | Without Vertigo; Placebo - Rizatriptan | With Vertigo; Rizatriptan - Placebo | Without Vertigo; Rizatriptan - Placebo
Started | 6 | 8 | 6 | 6
Completed | 6 | 7 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Twenty seven subjects completed screening tests and met study criteria. Twenty five of the 27 subjects enrolled completed both experimental study visits.
Groups:
- All Study Participants: Includes participants (migraineurs) with and without vertigo
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Motion Sickness to Post Vestibular Stimulus
Description: Scores are based on a scale developed by Graybiel which rates seven subjective and objective signs of motion sickness. The total scores ranged from from 0 to 25. Zero indicating no motion sickness. Greater than 16 indicates severe motion sickness. Trials were stopped if scores were 16 or greater. Scores were taken before and after each rotation.
Time Frame: Pre and Post Stimulus (about 6 minutes apart)
Population: Ten of the 25 subjects who completed both experimental visits developed negligible motion sickness induced by the stimulus following pre-medication with placebo. These data were not analyzed. It was posited that the presence/absence of vertigo would not impact the analysis of this outcome. The groups were combined for the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Rizatriptan Visit: Subjects were pre-treated with Rizatriptan prior to vestibular stimulation.
- Placebo Visit: Participants were pre-treated with placebo prior to vestibular stimulation.
Arm/Group | Rizatriptan Visit | Placebo Visit
Number analyzed (Participants) | 15 | 15
units on a scale | 5.1 [2 to 10] | 9 [4.9 to 10.9]
Statistical Analysis 1: Comparison: Rizatriptan Visit vs Placebo Visit; Test type: Superiority or Other; p = 0.007, Sign test

2. Secondary Outcome: Change From Baseline in Subjective Units of Distress to Post Vestibular Stimulus
Description: Subjective report of distress ranging from 0 to 10 based on the method of Wolpe. Zero indicates no distress and 10 indicates severe distress. Measures used in this analysis match the times used in the analysis for Outcome 1.
Time Frame: Pre and Post Stimulus (6 minutes apart)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Rizatriptan Visit | Placebo Visit
Number analyzed (Participants) | 15 | 15
units on a scale | 3 [0 to 5] | 2 [1 to 4]
Statistical Analysis 1: Comparison: Rizatriptan Visit vs Placebo Visit; Test type: Superiority or Other; p = .549, Sign test

ADVERSE EVENTS:
Time Frame: For the duration of the study visit.
Groups:
- Without Vertigo; Placebo: These participants suffered from migraines but did not have associated dizziness/vertigo. They received Placebo on one of the visits.
- Without Vertigo; Rizatriptan: These participants suffered from migraines but did not have associated dizziness/vertigo. They received Rizatriptan on one of the visits.
- With Vertigo; Placebo: These participants suffered from migraines with associated dizziness/vertigo. They received Placebo on one of the visits.
- With Vertigo; Rizatriptan: These participants suffered from migraines with associated dizziness/vertigo. They received Rizatriptan on one of the visits.
Arm/Group | Without Vertigo; Placebo | Without Vertigo; Rizatriptan | With Vertigo; Placebo | With Vertigo; Rizatriptan
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 1/14 | 0/14 | 0/12 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Without Vertigo; Placebo (N=14) | Without Vertigo; Rizatriptan (N=14) | With Vertigo; Placebo (N=12) | With Vertigo; Rizatriptan (N=13)
Increased Blood Pressure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On first experimental visit - Subject had an increase in blood pressure within the 2 hour window between taking pill and the rotational trials.
Nausea (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — On experimental visit one, the subject reported feeling nausea after taking the drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No